CLINICAL TRIAL: NCT04260997
Title: A Randomised, Double-Blinded, Parallel, Placebo-Controlled Study Investigating the Effect of a Probiotic, Lactobacillus Gasseri BNR17, on Body Composition and Weight Management in Overweight Adults.
Brief Title: Effect of a Probiotic, Lactobacillus Gasseri BNR17, on Body Composition and Weight Management in Overweight Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UAS Labs LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFCRO-112
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Weight Management

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Probiotic Product (Experimental)
  Interventions: Dietary Supplement: Lactobacillus gasseri BNR17™ capsule
- Placebo product (Placebo Comparator)
  Interventions: Other: Placebo capsule

INTERVENTIONS:
Dietary Supplement: Lactobacillus gasseri BNR17™ capsule — Once per day (QD), 12 weeks
  Arms: Oral Probiotic Product
Other: Placebo capsule — Once per day (QD), 12 weeks
  Arms: Placebo product

SUMMARY:
Lactobacillus gasseri BNR17™ has shown promise in several pre-clinical and randomized controlled clinical trials for weight management outcomes. The current randomized, double-blind, placebo-controlled, parallel-arm trial will further assess L. gasseri BNR17™ on body composition and weight management, and in a study population that is distinct to prior randomized controlled trials on the strain. The study will recruit 126 overweight adult participants who will be randomly assigned to consume L. gasseri BNR17™ or placebo once daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent;
* Aged between 25 and 65 years inclusive;
* Body mass index between 25.0 to 29.9 Kg/m2, inclusive;
* Waist-hip ratio of ≥0.91 for males and ≥0.81 for females;
* Sedentary lifestyle, exercising ≤2 times/week;
* Good general health, as determined by the investigator;
* Willing to consume the investigational product daily for the duration of the study;
* Outside the healthy parameters of visceral adipose tissue, defined as 762 cm3 for males and 256 cm3 for females.

Exclusion Criteria:

* Females who are pregnant, lactating or wish to become pregnant during the study;
* Participant regularly takes probiotic supplements, or has within the 4-weeks prior to randomisation or plans to during the study;
* Participant is hypersensitive to any of the components of the investigational product;
* Participant is severely immuno-compromised (HIV positive, transplant patient, on antirejection medications, on a steroid for >30 days, or has underwent chemotherapy or radiotherapy within the last year);
* Participant has Type 1 or Type 2 Diabetes Mellitus;
* Participant has a history of bariatric surgery;
* Participant has taken anti-obesity medication or supplements in the 12-weeks prior to randomisation or plans to during the study;
* Participant is actively or has recently (3 months prior to randomisation) participated in a weight loss program or weight change of 3 kg during the past 3 months;
* Participant has a life-threatening illness;
* Participant is on a glucose lowering medication, anti-psychotic drugs or any medication that the investigator determines could impact the results of the study; participant has commenced use, within 3-months of randomisation, anti-hypertensive drugs, anti-depressive drugs, statin or any other medication that the investigator determines could impact the results of the study;
* Participant has a history of co-existing gastrointestinal, and/or gynecological, and/or urologic pathology (e.g. colon cancer, colitis, Crohn's Disease, Celiac, Endometriosis, prostate cancer) or lactose intolerance;
* Participant has a recent history of drug and/or alcohol abuse at the time of enrolment;
* Participant is currently, or planning to participate in another study during the study period;
* Participant has a history of non-compliance;
* Participant has taken antibiotics in the 12-weeks prior to randomisation.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline to week 12 in visceral adipose tissue (VAT) | 12 weeks
  VAT will be assessed using dual energy x-ray absorptiometry

SECONDARY OUTCOMES:
Absolute change from baseline to week 12 in total fat mass | 12 weeks
Absolute change from baseline to week 12 in total lean mass | 12 weeks
Absolute change from baseline to week 12 in body weight | 12 weeks
Absolute change from baseline to week 12 in waist circumference | 12 weeks
Absolute change from baseline to week 12 in waist-to-hip ratio | 12 weeks
Absolute change from baseline to week 12 in blood glucose | 12 weeks
Absolute change from baseline to week 12 in HbA1c | 12 weeks
Absolute change from baseline to week 12 in blood insulin | 12 weeks
Absolute change from baseline to week 12 in hs-CRP | 12 weeks

OTHER OUTCOMES:
Gastrointestinal symptom rating scale | 12 weeks
Safety blood profile (clinical chemistry and full blood count) | 12 weeks
Vitals (systolic blood pressure, diastolic blood pressure, heart rate and temperature) | 12 weeks
Adverse events (frequency, severity and relatedness) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantia Food Clinical Trials, Cork, Ireland